CLINICAL TRIAL: NCT01676662
Title: An Evaluation of the Solace Bladder Control System in the Treatment of Female Subjects With Stress Urinary Incontinence
Brief Title: Solace European Confirmatory Trial
Acronym: SOLECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solace Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CD 1004
Record Dates: First submitted 2012-08-23; First posted 2012-08-31 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence; Urinary Incontinence, Stress; Urination Disorders; Urologic Diseases; Urological Manifestations; Signs and Symptoms
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Urination Disorders; Urologic Diseases; Urological Manifestations; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment on Day 0 (Experimental): Subjects who are treated with the Solace Bladder Control System upon entry into the trial.
  Interventions: Device: Solace Bladder Control System
- Sham Treatment on Day 0 (Sham Comparator): Patients who undergo a sham procedure upon entry into the trial, with treatment with the Solace Bladder Control System at 3 months after the sham procedure.
  Interventions: Device: Solace Bladder Control System; Device: Solace Sham Treatment

INTERVENTIONS:
Device: Solace Bladder Control System — Subjects may undergo treatment every 12 months until study completion.
Device: Solace Sham Treatment — Sham procedure that resembles treatment with the Solace Bladder Control System
  Arms: Sham Treatment on Day 0

SUMMARY:
The Solace European Confirmatory (SOLECT) Trial is designed to determine whether the Solace Bladder Control System is safe and effective for the treatment of Stress Urinary Incontinence (SUI) in adult females.

DETAILED DESCRIPTION:
Subject will undergo treatment with the Solace Bladder Control System or a sham procedure, with the results being compared at 3 months.

All patients undergoing sham treatment are treated at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years of age or older with stress urinary incontinence (SUI)
* Experienced SUI for at least 12 months and attempted and failed prior noninvasive treatment
* Willing to undergo cystoscopic procedures required and 36 month follow-up
* On stable medication for a minimum of 3 months
* Free of local genital skin infection
* Positive Pad Weight Test
* Free of impassable urethral strictures, trauma or necrosis

Exclusion Criteria (must answer NO):

* Pregnant or planning to become pregnant during the study period
* Non-ambulatory or bedridden or physically unable to complete test exercises
* Morbidly obese (defined as BMI ≥ 40 kg/m2)
* Bladder infection (including bladder inflammation or edema) or UTI within 3 months
* History of recurrent urinary tract infections
* Prior surgical procedure for incontinence within the past 6 months
* Is taking medications for urinary incontinence other than anticholinergics
* History of kidney stones
* Has a prosthetic heart valve
* Unable to tolerate any form of antibiotic
* Taking anticoagulation therapy, other than aspirin
* Has urinary incontinence due to Intrinsic Sphincter Deficiency (ISD)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of life as assessed by pad weight tests assessments and questionnaires | 3 Months
  Comparison of increases in pad weight test and patient reported outcomes on questionnaires.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | 3 Months
  Site-reported adverse events designated as related to the treatment.
Severity of treatment-related adverse events | 3 Months
  Site-reported adverse events designated as related to the treatment.

OTHER OUTCOMES:
Incidence of all adverse events | 36 Months
  Rate of incidence of all adverse events for all patients
Improvement in quality of life in all patients assessed with pad weight tests and questionnaires | 36 Months
Severity of all adverse events | 36 Months
  Severity of all adverse events for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Tommaselli, M.D., Principal Investigator — University of Naples
Locations (7):
- Belgium (3):
  - University of Antwerp Hospital (Universitair Ziekenhuis Antwerpen), Antwerp, Edegem
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
- Italy (2):
  - University of Naples (Università Degli Studi Di Napoli "Federico II" ), Naples (Napoli)
  - Universita Campus Bio-medico di Roma, Rome
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht University Medical Center, Maastricht

IPD SHARING:
Plan to Share IPD: No
Pending publication of results

REFERENCES:
- [Result] Wyndaele JJ, De Wachter S, Tommaselli GA, Angioli R, de Wildt MJ, Everaert KC, Michielsen DP, Van Koeveringe GA. A randomized, controlled clinical trial of an intravesical pressure-attenuation balloon system for the treatment of stress urinary incontinence in females. Neurourol Urodyn. 2016 Feb;35(2):252-9. doi: 10.1002/nau.22708. Epub 2015 Jan 16. PMID 25598453